CLINICAL TRIAL: NCT00697840
Title: Study to Assess the Safety, Immunogenicity and Reactogenicity of GSK Biologicals' (Previously SmithKline Beecham Biologicals') Adjuvanted Recombinant Hepatitis B Vaccine, Recombinant Hepatitis B Vaccine New Formulation and Engerix™-B
Brief Title: Safety, Immunogenicity and Reactogenicity of Recombinant Hepatitis B Vaccine (Adjuvanted & New Formulation) and Engerix™-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208129/019
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant hepatitis B vaccine; Adjuvant
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL 208129
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B
- Group C (Experimental)
  Interventions: Biological: Vaccine containing HBsAg absorbed on aluminium salts - experimental formulation

INTERVENTIONS:
Biological: Engerix™-B — Intramuscular injection, 2 doses
  Arms: Group B
Biological: HBV-MPL 208129 — Intramuscular injection, 2 doses
  Arms: Group A
Biological: Vaccine containing HBsAg absorbed on aluminium salts - experimental formulation — Intramuscular injection, 2 doses; experimental formulation
  Arms: Group C

SUMMARY:
The purpose of the present trial is to assess the safety, reactogenicity and immunogenicity of adjuvanted hepatitis B vaccine, Engerix™-B and hepatitis B vaccine new formulation when administered at 0, 6 months

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years old.
* Written informed consent will have been obtained from the subjects.
* Good physical condition as established by physical examination and history taking at the time of entry.
* Female participants will avoid becoming pregnant during the study period and they will have been on a contraceptive program for at least 2 months before entry

Exclusion Criteria:

* Pregnancy or lactation.
* Positive titres for anti HBs antibody.
* Any vaccination against hepatitis B in the past.
* Any previous administration of MPL.
* Elevated serum liver enzymes.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Axillary temperature > 37.5°C at the time of injection.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Any treatment with immunosuppressive or immunostimulant therapy.
* Any chronic drug treatment, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Simultaneous administration of any other vaccine(s).
* Administration of any immunoglobulin during the study period.
* Simultaneous participation in any other clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 1995-06; Primary Completion 1996-01 (Actual); Study Completion 1996-01 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At month 7
Occurrence and intensity of solicited local and general symptoms | 4-day follow-up after vaccination
Occurrence of unsolicited adverse events | 30-days after vaccination
Incidence of serious adverse events | Throughout the study period
Anti-Hbs antibody concentrations | Months 1, 6 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Vienna, Austria